CLINICAL TRIAL: NCT06174363
Title: Analgesic Efficacy of Maxigesic Added to Opioid Based-PCA in Patients Undergoing Breast Cancer Surgery
Brief Title: Analgesic Efficacy of Maxigesic in Breast Cancer Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Jin Sun Cho, M.D, PhD, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 4-2022-1650
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Control group: 0.9% saline solution/ Study group: Maxigesic
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Placebo Comparator): Group administered Maxigesic solution
  Interventions: Drug: Maxigesic
- Control group (Experimental): Group administerd 0.9% saline solution
  Interventions: Drug: 0.9% saline solution

INTERVENTIONS:
Drug: Maxigesic — For postoperative analgesia, 50 mcg of fentanyl was administered 15 minutes before the end of surgery, and IV-PCA (fentanyl 1.0 mcg/kg, ramosetron 0.3 mg, total 250cc, infusion rate 5cc/h, bolus 0.5 cc, lock-out time 15min) is started. Additionally, in the Maxigesic group, one vial of Maxigesic (acetaminophen 1000mg/ ibuprofen 300mg) is administered 15 minutes before the end of the surgery, and 2 vials of Maxigesic are added to the IV-PCA.
  Arms: Study group
Drug: 0.9% saline solution — For postoperative analgesia, 50 mcg of fentanyl was administered 15 minutes before the end of surgery, and IV-PCA (fentanyl 1.0 mcg/kg, ramosetron 0.3 mg, total 250cc, infusion rate 5cc/h, bolus 0.5 cc, lock-out time 15min) is started. Additionally, in the control group, the same amount of 0.9% saline solution with Maxigesic is administered.
  Arms: Control group

SUMMARY:
The present study aims to find a perioperative analgesic method that provides sufficient analgesia while reducing immune compromise in cancer surgery. This study is to investigate the analgesic effect and safety of Maxigesic inj. (a combination of acetaminophen 1000 mg and ibuprofen 300 mg), which is added to opioid-based IV-PCA in patients undergoing breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 20 to 70 years with ASA classification 1 to 3 undergoing breast cancer surgery (cancer resection or reconstruction)

Exclusion Criteria:

* ASA classification 4/ allergy to acetaminophen, NSAIDs, opioid/ severe liver or renal dysfunction/ pregnancy

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-12-28 (Actual); Primary Completion 2025-12-26 (Estimated); Study Completion 2025-12-26 (Estimated)

PRIMARY OUTCOMES:
Analgesic effect of Maxigesic | postoperative 30 minutes/ 6 hours/ 24 hours/ 48 hours
  Postoperative pain intensity is assessed with NRS: numerical rating scales (0 = no pain ∼ 10 = worst pain).

SECONDARY OUTCOMES:
Incidence of Adverse reactions (Safety) | postoperative 30 minutes/ 6 hours/ 24 hours/ 48 hours
  Adverse reactions related to NSAIDs: headache, dizziness, nausea, vomiting, itching, drowsiness, abdominal pain, constipation, gastrointestinal bleeding, hypotension.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Data obtained through this study may be provided to qualified researchers with an academic interest in perioperative analgesia in cancer surgery. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.